CLINICAL TRIAL: NCT05183360
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Dose and Multiple Rising Oral Doses of BI 706321 in Healthy Japanese Male Subjects and Single Oral Dose of BI 706321 in Healthy Chinese Male Subjects (Double-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study in Healthy Japanese and Chinese Men to Test How Well Different Doses of BI 706321 Are Tolerated
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1425-0008
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Results first posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo Matching BI 706321 (Part I) (Placebo Comparator): This trial consisted of two parts: a single-dose part and a multiple-dose part.
  Single-Dose Part:
  On Day 1, after fasting for at least 10 hours overnight, participants received a single dose of placebo tablets matching BI 706321.
  Multiple-Dose Part:
  From Day 6 to Day 19, after fasting for at least 10 hours overnight, participants received a daily dose of placebo tablets matching BI 706321.
  Interventions: Drug: Placebo
- 2 mg BI 706321 (Part I) (Experimental): This trial consisted of two parts: a single-dose part and a multiple-dose part.
  Single-Dose Part:
  On Day 1, after fasting for at least 10 hours overnight, participants received a single dose of one 2 milligrams (mg) tablet BI 706321.
  Multiple-Dose Part:
  From Day 6 to Day 19, after fasting for at least 10 hours overnight, participants received a daily dose of one 2 mg tablet BI 706321.
  Interventions: Drug: BI 706321
- 5 mg BI 706321 (Part I) (Experimental): This trial consisted of two parts: a single-dose part and a multiple-dose part.
  Single-Dose Part:
  On Day 1, after fasting for at least 10 hours overnight, participants received a single dose of one 5 mg tablet BI 706321.
  Multiple-Dose Part:
  From Day 6 to Day 19, after fasting for at least 10 hours overnight, participants received a daily dose of one 5 mg tablet BI 706321.
  Interventions: Drug: BI 706321
- 8 mg BI 706321 (Part I) (Experimental): This trial consisted of two parts: a single-dose part and a multiple-dose part.
  Single-Dose Part:
  On Day 1, after fasting for at least 10 hours overnight, participants received a single dose of three tablets totaling 8 mg of BI 706321.
  Multiple-Dose Part:
  From Day 6 to Day 19, after fasting for at least 10 hours overnight, participants received a daily dose of three tablets totaling 8 mg of BI 706321.
  Interventions: Drug: BI 706321
- 10 mg BI 706321 (Part I) (Experimental): This trial consisted of two parts: a single-dose part and a multiple-dose part.
  Single-Dose Part:
  On Day 1, after fasting for at least 10 hours overnight, participants received a single dose of two tablets totaling 10 mg of BI 706321.
  Multiple-Dose Part:
  From Day 6 to Day 19, after fasting for at least 10 hours overnight, participants received a daily dose of two tablets totaling 10 mg of BI 706321.
  Interventions: Drug: BI 706321

INTERVENTIONS:
Drug: BI 706321 — BI 706321, tablet, oral use
  Arms: 10 mg BI 706321 (Part I); 2 mg BI 706321 (Part I); 5 mg BI 706321 (Part I); 8 mg BI 706321 (Part I)
Drug: Placebo — Placebo, tablet, oral use
  Arms: Placebo Matching BI 706321 (Part I)

SUMMARY:
Part I: The main objectives of this trial are to investigate safety, tolerability, and pharmacokinetics (PK) of BI 706321 in healthy Japanese male subjects following oral administration of multiple rising doses.

Part II: The main objectives of this trial are to investigate safety, tolerability, and pharmacokinetics (PK) of BI 706321 in healthy Chinese male subjects following oral administration of single dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure [BP], pulse rate (PR) including body temperature, 12-lead electrocardiogram (ECG), and clinical laboratory tests at screening visit
* Part I: Japanese ethnicity, according to the following criteria:

  -- born in Japan, have lived outside of Japan <10 years
* Part II: Chinese ethnicity including Taiwanese, according to the following criteria:

  -- have parents and grandparents who are Chinese
* Age of 20 to 45 years (inclusive) at screening visit
* Body mass index (BMI) of 18.5 to 25.0kg/m2 (inclusive) at screening visit
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Willingness to comply with contraception requirements. Subjects who are sexually active must use adequate contraception methods throughout the trial and until three months after the last administration of trial medication. Adequate methods are:

  * A vasectomy performed at least 1 year prior to screening and with medical assessment of the surgical success or
  * Surgical sterilization, including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy, of the subject's female partner or
  * The use of condoms, if the female partner uses an adequate contraception method in addition, e.g., intrauterine device (IUD), or hormonal contraception, such as implants and injectables, combined with oral or vaginal contraceptives, that started at least 2 months prior to first drug administration, or barrier method, e.g., diaphragm with spermicide

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR, body temperature or ECG) deviating from normal and assessed as clinically relevant by the investigator at screening visit
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 40 to 90 mmHg, or pulse rate outside the range of 40 to 99 bpm at screening visit
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance at screening visit
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders, per investigator judgement
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, placebo-controlled, double-blind trial conducted in two parts. Part I involved 48 healthy Japanese males who received BI 706321 as single and multiple rising doses. Part II was planned to involve healthy Chinese males receiving a single dose of BI 706321, but the trial was prematurely discontinued before starting Part II, and no participants were enrolled in Part II.
Pre-assignment Details: 48 Japanese male participants who met all inclusion criteria and no exclusion criteria were enrolled in Part I of the trial. All received the trial medication and placebo as planned and completed the trial per protocol. Participants were free to withdraw at any time and were closely monitored. The trial was prematurely discontinued per protocol before Part II began.
Period: Overall Study
Arm/Group | Placebo Matching BI 706321 (Part I) | 2 mg BI 706321 (Part I) | 5 mg BI 706321 (Part I) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I)
Started | 12 | 9 | 9 | 9 | 9
Completed | 12 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: all participants who were randomized and treated with at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching BI 706321 (Part I) | 2 mg BI 706321 (Part I) | 5 mg BI 706321 (Part I) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I) | Total
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.8 (7.9) | 31.9 (8.2) | 29.4 (7.6) | 31.9 (7.5) | 32.3 (6.5) | 31.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 9 | 9 | 9 | 9 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 9 | 9 | 9 | 9 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 9 | 9 | 9 | 9 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events
Description: The percentage of participants treated with investigational drug who experience such an event.
  Percentage of participants with treatment-emergent adverse events assessed as drug-related by the investigator are reported.
  Percentages are calculated using total number of participants per treatment as the denominator.
Time Frame: From 1st drug administration on Day 1 till Day 19 + 16 days Residual Effect Period (REP), up to 35 days.
Population: Treated set: all participants who were randomized and treated with at least one dose of the study drug.
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Placebo Matching BI 706321 (Part I) | 2 mg BI 706321 (Part I) | 5 mg BI 706321 (Part I) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
Percentage (%) of participants | 8.3 | 11.1 | 44.4 | 66.7 | 88.9

2. Secondary Outcome: Single-Dose Part: Area Under the Concentration-time Curve of the BI 706321 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUCR0-∞)
Description: The area under the concentration-time curve of the BI 706321 in plasma over the time interval from 0 extrapolated to infinity (AUCR0-∞) after the first dose administration is reported.
Time Frame: Within 3 hours prior to administration and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours, and 1.5, 2, 3, and 4 days after first BI 706321 administration.
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all participants in the treated set (TS) who provide at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*(nanomoles/L)
Groups:
- 2 mg BI 706321 (Part I - Single-Dose Part Only): Single-Dose Part:
  On Day 1, after fasting for at least 10 hours overnight, participants received a single dose of one 2 milligrams (mg) tablet BI 706321.
- 5 mg BI 706321 (Part I - Single-Dose Part Only): Single-Dose Part:
  On Day 1, after fasting for at least 10 hours overnight, participants received a single dose of one 5 mg tablet BI 706321.
- 8 mg BI 706321 (Part I): Single-Dose Part:
  On Day 1, after fasting for at least 10 hours overnight, participants received a single dose of three tablets totaling 8 mg of BI 706321.
- 10 mg BI 706321 (Part I - Single-Dose Part Only): Single-Dose Part:
  On Day 1, after fasting for at least 10 hours overnight, participants received a single dose of two tablets totaling 10 mg of BI 706321.
Arm/Group | 2 mg BI 706321 (Part I - Single-Dose Part Only) | 5 mg BI 706321 (Part I - Single-Dose Part Only) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I - Single-Dose Part Only)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Hours*(nanomoles/L) | 78.0 (31.8) | 196 (28.7) | 447 (32.9) | 393 (25.7)

3. Secondary Outcome: Single-Dose Part: Maximum Measured Concentration of BI 706321 in Plasma (Cmax)
Description: The maximum measured concentration of BI 706321 in plasma (Cmax) after the first dose administration is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per Liters
Arm/Group | 2 mg BI 706321 (Part I - Single-Dose Part Only) | 5 mg BI 706321 (Part I - Single-Dose Part Only) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I - Single-Dose Part Only)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Nanomoles per Liters | 3.00 (30.6) | 8.20 (47.9) | 18.4 (35.4) | 17.7 (36.4)

4. Secondary Outcome: Single-Dose Part: Time From Dosing to Maximum Measured Concentration of BI 706321 in Plasma
Description: The time from dosing to maximum measured concentration of BI 706321 in plasma after first drug administration is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 2 mg BI 706321 (Part I - Single-Dose Part Only) | 5 mg BI 706321 (Part I - Single-Dose Part Only) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I - Single-Dose Part Only)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Hours | 5.00 [2.00 to 5.00] | 5.00 [2.00 to 5.00] | 5.00 [2.00 to 5.00] | 5.00 [2.00 to 6.00]

5. Secondary Outcome: Area Under the Concentration-time Curve of BI 706321 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ,ss)
Description: Area under the concentration-time curve of BI 706321 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) after single and multiple dose administration is reported.
Time Frame: Within 3 hours prior to administration and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours, and 1.5, 2, 3, and 4 days, and additional time points up to 26 days after first BI 706321 administration.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*(nanomoles/L)
Arm/Group | 2 mg BI 706321 (Part I) | 5 mg BI 706321 (Part I) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Hours*(nanomoles/L) | 144 (44.8) | 297 (21.9) | 764 (19.3) | 641 (23.0)

6. Secondary Outcome: Maximum Measured Concentration of BI 706321 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss)
Description: Maximum measured concentration of BI 706321 in plasma at steady state over a uniform dosing interval τ (Cmax,ss) after single and multiple dose administration is reported
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per Liters
Arm/Group | 2 mg BI 706321 (Part I) | 5 mg BI 706321 (Part I) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Nanomoles per Liters | 7.30 (55.4) | 20.0 (25.7) | 52.4 (11.1) | 43.3 (24.5)

7. Secondary Outcome: Minimum Concentration of BI 706321 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmin,ss)
Description: Minimum concentration of BI 706321 in plasma at steady state over a uniform dosing interval τ (Cmin,ss) after single and multiple dose administration is reported.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per Liters
Arm/Group | 2 mg BI 706321 (Part I) | 5 mg BI 706321 (Part I) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Nanomoles per Liters | 3.47 (39.0) | 7.88 (31.9) | 20.8 (27.0) | 17.4 (25.1)

8. Secondary Outcome: Accumulation Ratio Based on Cₘₐₓ (Rᴀ,ᴄₘₐₓ,ₛₛ)
Description: The accumulation ratio based on Cₘₐₓ (Rᴀ,ᴄₘₐₓ,ₛₛ) shows how much the drug concentration increases at steady state compared to the first dose. It is calculated as a ratio of Cₘₐₓ at steady state (Cₘₐₓ,ₛₛ) and Cₘₐₓ after the first dose (Cₘₐₓ).
  Rᴀ,ᴄₘₐₓ,ₛₛ = Cₘₐₓₛₛ/Cₘₐₓ.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio - no unit
Arm/Group | 2 mg BI 706321 (Part I) | 5 mg BI 706321 (Part I) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Ratio - no unit | 2.43 (34.5) | 2.44 (25.2) | 2.85 (36.2) | 2.44 (23.1)

9. Secondary Outcome: Accumulation Ratio Based on AUC₀-ₜ (Rᴀ,ᴀᴜᴄ₀-ₜ,ₛₛ)
Description: The accumulation ratio based on AUC₀-ₜ (Rᴀ,ᴀᴜᴄ₀-ₜ,ₛₛ) shows how much the total drug exposure over a uniform dosing interval τ increases at steady state compared to the first dose. It is calculated as a ration of AUC₀-ₜ at steady state (AUC₀-ₜₛₛ) and AUC₀-ₜ after the first dose (AUC₀-ₜ).
  Rᴀ,ᴀᴜᴄ₀-ₜ,ₛₛ = AUC₀-ₜₛₛ/AUC₀-ₜ.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio - no unit
Arm/Group | 2 mg BI 706321 (Part I) | 5 mg BI 706321 (Part I) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Ratio - no unit | 3.03 (29.1) | 3.00 (23.2) | 3.52 (31.0) | 3.12 (18.9)

ADVERSE EVENTS:
Time Frame: Adverse Events and All-Cause Mortality: From 1st drug administration on Day 1 till Day 19 + 16 days (REP), up to 35 days
Description: Treated set: all participants who were randomized and treated with at least one dose of the study drug.
Arm/Group | Placebo Matching BI 706321 (Part I) | 2 mg BI 706321 (Part I) | 5 mg BI 706321 (Part I) | 8 mg BI 706321 (Part I) | 10 mg BI 706321 (Part I)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 5/12 | 2/9 | 5/9 | 6/9 | 8/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 706321 (Part I) (N=12) | 2 mg BI 706321 (Part I) (N=9) | 5 mg BI 706321 (Part I) (N=9) | 8 mg BI 706321 (Part I) (N=9) | 10 mg BI 706321 (Part I) (N=9)
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 2 | 5 | 7
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 2 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 1 | 3
Headache (Nervous system disorders) | 1 | 1 | 2 | 4 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The trial was prematurely discontinued per protocol before Part II began.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT05183360/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT05183360/SAP_001.pdf